CLINICAL TRIAL: NCT02582619
Title: Development of a Multidisciplinary Model to Guide Employment Outcomes in People Living With Spinal Cord Injuries in South Africa.
Brief Title: Multidisciplinary Model to Guide Employment Amongst PLWSCI
Status: Completed | Type: Observational
Sponsor: University of KwaZulu (Other)
Responsible Party: Principal Investigator, Ntsikelelo Pefile, Mr, University of KwaZulu
Other Study IDs: BE499/14
Record Dates: First submitted 2015-10-15; First posted 2015-10-21 (Estimated); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Spinal Cord Injury
Keywords: Spinal Cord Injury and Employment
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Focus Groups

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Rehabilitation Professionals: Focus group consisting of rehabilitation professionals that will inform the study on vocational rehabilitation interventions rendered during acute to in-patient rehabilitation in KwaZulu-Natal.
  Interventions: Other: Focus groups, semistructured interviews and Delphi rounds
- People living with Spinal Cord Injuries (PLWSCI): Focus group consisting of PLWSCI that will inform the study on the perspective of the patient on vocational rehabilitation needs or desires during acute care and in-patient rehabilitation.
  This group will inform the study on the employment rate amongst people living with spinal cord injuries as well as factors that influence employment.
  This group will also inform the study on the perceived barriers and facilitators of employment
  Interventions: Other: Focus groups, semistructured interviews and Delphi rounds
- Stakeholders: Representatives from the following departments or organisations will be invited to participate in the interviews and focus groups:
  Government Departments:
  Education Social Development Health Labour Transport
  Private Companies:
  Insurance Companies and Health Risk Management companies Non-profit Organisations QASA DPSA
  Interventions: Other: Focus groups, semistructured interviews and Delphi rounds
- Experts: A delphi technique will be used to get an expert opinion and consensus on the aspects of the model to be developed.
  Interventions: Other: Focus groups, semistructured interviews and Delphi rounds

INTERVENTIONS:
Other: Focus groups, semistructured interviews and Delphi rounds

SUMMARY:
Spinal cord injury often results in complete or partial loss of functioning of the upper and or lower limbs, leading to the affected individual experiencing difficulties in performing activities of daily living. This in turn results in reduced participation in social, religious, recreational and economic activities (employment). Globally, there is a low employment rate (11-67%) amongst PLWSCI. In South Africa, according to Statistics South Africa, the unemployment rate of people with disabilities is estimated to be 25.2%. However, there is no information available on employment amongst PLWSCI in South Africa.

Furthermore, there is insufficient knowledge related to SCI in South Africa to enable a model to be developed and implemented. Data on the current SCI rehabilitation practices (with specific reference to vocational rehabilitation); employment status and factors (both personal and environmental); barriers and facilitators of employment amongst PLWSCI is limited. This information is needed to develop a return to work model for individuals with SCI in South Africa.

In South Africa, a legal framework exists that promotes the employment as well as assistance of people with disabilities in the workplace, such as: the Constitution of Republic of South Africa, 1996; the Employment Equity Act (EEA), 1998; the Promotion of Equality and Prevention of Unfair Discrimination Act (PEPUDA), 2000; Labour Relations Act (LRA), 1995; Skills Development Act (SDA), 1998; Public Service Act (PSA), 1994; Basic Conditions of Employment Act (BCEA), 1997 and the Integrated National Disability Strategy (2000). However, rehabilitation interventions provided in rehabilitation institutions are mainly medical, with limited attempts to prepare those with SCI to return to gainful employment. There is therefore a need for a well-coordinated, multi-sectorial, multi-disciplinary and multi-factorial rehabilitation intervention that will promote the employment of PLWSCI in South Africa.

DETAILED DESCRIPTION:
This is a cross-sectional study in which mixed methods will be used in various phases of the study. Mixed methods involve the collection and analysis of both quantitative and qualitative data in a single study. Data are collected concurrently or sequentially and integrated at one or more stages during the research process. This study will be divided into 3 phases with stages to answer the objectives.

Phase one of this study will attempt to answer objectives 1-3 of the study. Stage 1 will include a systematic review of literature to identify the most effective vocational rehabilitation interventions amongst PLWSCI. Stage 2 will determine rehabilitation services rendered to individual who sustain SCI in South Africa with an intention of identifying gaps in vocational rehabilitation practices by retrospectively analysing medical files. This phase will be concluded by a focus group to further explore current vocational rehabilitation practices rendered to PLWSCI (Stage3).

Phase two will answer objectives 4-5. Stage 1 of this phase will determine the employment status as well as factors that influence employment amongst PLWSCI. Stage 2 will determine the barriers and facilitators of employment amongst PLWSCI. Results obtained from phase 1 to 2, will be utilised to by the researcher to develop the proposed model.

The final phase will aim to develop, validate and refine the model. Stage 1 of this phase will include the researcher using the information gained in previous phases to develop the proposed model. The second stage will include a focus group to validate the content of the proposed model. The last stage will included obtaining consensus amongst the stakeholders regarding the structure and the content of the proposed model and subsequently refine it.

ELIGIBILITY:
Phase One:

Inclusion Criteria:

• Rehabilitation professionals who are directly involved in the management of individuals who sustain SCI and have more than 1 year of working experience post community service.

Exclusion Criteria:

• Rehabilitation professionals who are not directly involved in the management of individuals who sustain SCI and have less than 1 year working experience post community service.

Phase Two :

Inclusion Criteria:

• Person who sustained injury to the spine, resulting in permanent neurological damage (complete or incomplete) and must reside in a rural, peri-urban and urban.

Exclusion Criteria

• People living with spinal cord injuries who cannot verbally communicate

Phase Three Inclusion Criteria

* PLWSCI Injury to who resides in a rural, peri-urban and urban.
* Rehabilitation professionals who are directly involved in the management of individuals who sustain SCI and have more than 2 years of experience post community service.
* An individual who is full time employed in a supervisory and managerial capacity in both private and public sector, currently have subordinates who are PLWSCI.
* A representative from the Disability Section of an insurance company that is the member of the LOA.

Exclusion Criteria

* PLWSCI who cannot verbally communicate.
* Rehabilitation professionals who are not directly involved in the management of individuals who sustain SCI and have less than two years of experience post community service.
* An individual who is employed on a part-time basis and not in supervisory or managerial positions and have no subordinates who are PLWSCI.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Phase One :
  Rehabilitation Professionals People living with Spinal Cord Injuries Representatives from various working environment
Sampling Method: Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2019-08 (Actual); Study Completion 2021-08 (Actual)

PRIMARY OUTCOMES:
A multidisciplinary model to guide employment amongst people living with spinal cord injuries | 18 months
  The final model will be developed using all the information gained from the Phase one and two of the study. A validation process will be done through the delphi rounds.

SECONDARY OUTCOMES:
Systematic Review of effective Vocational Rehabilitation interventions amongst People Living With Spinal Cord Injuries | Five Months
  The review study will follow the Chocrane A journal article will be published in a peer reviewed journal.
Rehabilitation Practices that promote employability of People Living with Spinal Cord Injuries | Three months
  Stage 2 and Stage Three of Phase one will develop a matrix or guideline of vocational rehabilitation interventions throughout the phases of rehabilitation.
Employment and Factors that affect employment amongst People living with Spinal Cord Injuries | Five months
  Employment rates and nature of employment will be quantified using the International Labour Organisation definition of employment. The Factors affecting employment will also be quantified using the modified Life Situation Questionnaire.
Barriers and Facilitators of employment amongst people living with spinal cord injuries. | 8 months
  Interviews and focus groups will be conducted to determine the barriers and facilitators of employment amongst PLWSCI.

CONTACTS AND LOCATIONS:
Overall Officials: Ntsikelelo Pefile, MScMedSc, Principal Investigator — University of KwaZulu
Locations (3):
- South Africa (3):
  - King Dinizulu Hospital, Durban, KwaZulu-Natal
  - Phoenix Spinal Rehabilitation Centre, Durban, KwaZulu-Natal
  - Greys Hospital, Pietermaritzburg, KwaZulu-Natal

REFERENCES:
- [Background] Anderson, D., Dumont, S., Azzaria, L., Le Bourdais, M., & Noreau, L. ( 2007). Determinants of return to work among spinal cord injury patients: A literature review. Journal of Vocational Rehabilitation , 27(1), 57-68.
- [Background] Bromley, I. (2006). Tetraplegia and Paraplegia. Sixth ed. London: Churchill Livingstone Elsevier.
- [Background] Catz A, Itzkovich M, Agranov E, Ring H, Tamir A. SCIM--spinal cord independence measure: a new disability scale for patients with spinal cord lesions. Spinal Cord. 1997 Dec;35(12):850-6. doi: 10.1038/sj.sc.3100504. PMID 9429264
- [Background] Chan SK, Man DW. Barriers to returning to work for people with spinal cord injuries: a focus group study. Work. 2005;25(4):325-32. PMID 16340109
- [Background] Coetzee, Z. G., C; van der Westhuizen, R; Van Niekerk, L. (2011). Re-conceptualising vocational rehabilitation services towards an inter-sectoral model. South African Journal of Occupational Therapy, 41(2), 32-36.
- [Background] Department of Health (South Africa). (2000). National Rehabilitation Policy. Pretoria: Government Printer.
- [Background] DeVivo M, Biering-Sorensen F, Charlifue S, Noonan V, Post M, Stripling T, Wing P; Executive Committee for the International SCI Data Sets Committees. International Spinal Cord Injury Core Data Set. Spinal Cord. 2006 Sep;44(9):535-40. doi: 10.1038/sj.sc.3101958. PMID 16955073
- [Background] DeVivo MJ, Biering-Sorensen F, New P, Chen Y; International Spinal Cord Injury Data Set. Standardization of data analysis and reporting of results from the International Spinal Cord Injury Core Data Set. Spinal Cord. 2011 May;49(5):596-9. doi: 10.1038/sc.2010.172. Epub 2010 Dec 7. PMID 21135863
- [Background] Dewbury,G., Clarke, K.,Randall, D., Rouncefield, M., Sommerville, I. (2004). The anti-social model of disability Disability and Society 19(2). 145-158.
- [Background] Domholdt, E. (2005). Rehabilitation Research: Principles and Applications. Third ed. Missouri: Elsevier Saunders.
- [Background] Dumont RJ, Okonkwo DO, Verma S, Hurlbert RJ, Boulos PT, Ellegala DB, Dumont AS. Acute spinal cord injury, part I: pathophysiologic mechanisms. Clin Neuropharmacol. 2001 Sep-Oct;24(5):254-64. doi: 10.1097/00002826-200109000-00002. PMID 11586110
- [Background] Ekong CE, Tator CH. Spinal cord injury in the work force. Can J Surg. 1985 Mar;28(2):165-7. PMID 3971241
- [Background] Escorpizo, R., Miller,W.C., Trenaman, L.M. (2012). Work and Employment Spinal Cord Rehabilitation Evidence, 4.0., 1-14.
- [Background] Fielingsdorf K, Dunn RN. Cervical spine injury outcome--a review of 101 cases treated in a tertiary referral unit. S Afr Med J. 2007 Mar;97(3):203-7. PMID 17440669
- [Background] Gobelet C, Luthi F, Al-Khodairy AT, Chamberlain MA. Vocational rehabilitation: a multidisciplinary intervention. Disabil Rehabil. 2007 Sep 15;29(17):1405-10. doi: 10.1080/09638280701315060. PMID 17729086
- [Background] Hallin P, Sullivan M, Kreuter M. Spinal cord injury and quality of life measures: a review of instrument psychometric quality. Spinal Cord. 2000 Sep;38(9):509-23. doi: 10.1038/sj.sc.3101054. PMID 11035471
- [Background] Hart C, Williams E. Epidemiology of spinal cord injuries: a reflection of changes in South African society. Paraplegia. 1994 Nov;32(11):709-14. doi: 10.1038/sc.1994.115. PMID 7885712
- [Background] Harvey, L. (2008). Management of Spinal Cord Injuries : A Guide for Physiotherapists. London: Butterworth Heinemann.
- [Background] Hess DR. Retrospective studies and chart reviews. Respir Care. 2004 Oct;49(10):1171-4. PMID 15447798
- [Background] Higgins, J.P.T., & Green, S. (2009). Cochrane Handbook for Systematic Reviews of Interventions England The Cochrane Collaboration and John Wiley & Sons (LTD).
- [Background] Hills, L.& Cullen, E. (2007). A study into the employment trends of individuals treated at a spinal cord injury centre. International Journal of Therapy and Rehabilitation, 14(8), 350-355.
- [Background] Hsu, C. S., BA. (2007). The Delphi Technique: Making Sense of Consesus. Practical Assessement Research and Evaluation, 12(10), 1-8.
- [Background] Itzkovich M, Gelernter I, Biering-Sorensen F, Weeks C, Laramee MT, Craven BC, Tonack M, Hitzig SL, Glaser E, Zeilig G, Aito S, Scivoletto G, Mecci M, Chadwick RJ, El Masry WS, Osman A, Glass CA, Silva P, Soni BM, Gardner BP, Savic G, Bergstrom EM, Bluvshtein V, Ronen J, Catz A. The Spinal Cord Independence Measure (SCIM) version III: reliability and validity in a multi-center international study. Disabil Rehabil. 2007 Dec 30;29(24):1926-33. doi: 10.1080/09638280601046302. Epub 2007 Mar 5. PMID 17852230
- [Background] Kidd PS, Parshall MB. Getting the focus and the group: enhancing analytical rigor in focus group research. Qual Health Res. 2000 May;10(3):293-308. doi: 10.1177/104973200129118453. PMID 10947477
- [Background] Krause JS, Sternberg M, Maides J, Lottes S. Employment after spinal cord injury: differences related to geographic region, gender, and race. Arch Phys Med Rehabil. 1998 Jun;79(6):615-24. doi: 10.1016/s0003-9993(98)90033-8. PMID 9630138
- [Background] Krause JS. Years to employment after spinal cord injury. Arch Phys Med Rehabil. 2003 Sep;84(9):1282-9. doi: 10.1016/s0003-9993(03)00265-x. PMID 13680562
- [Background] Krause JS, Carter RE, Pickelsimer EE, Wilson D. A prospective study of health and risk of mortality after spinal cord injury. Arch Phys Med Rehabil. 2008 Aug;89(8):1482-91. doi: 10.1016/j.apmr.2007.11.062. PMID 18674984
- [Background] Kroll T, Neri MT, Miller K. Using mixed methods in disability and rehabilitation research. Rehabil Nurs. 2005 May-Jun;30(3):106-13; discussion 113. doi: 10.1002/j.2048-7940.2005.tb00372.x. PMID 15912675
- [Background] Kroll T, Barbour R, Harris J. Using focus groups in disability research. Qual Health Res. 2007 May;17(5):690-8. doi: 10.1177/1049732307301488. PMID 17478650
- [Background] le Roux JC, Dunn RN. Gunshot injuries of the spine--a review of 49 cases managed at the Groote Schuur Acute Spinal Cord Injury Unit. S Afr J Surg. 2005 Nov;43(4):165-8. PMID 16440591
- [Background] Lidal IB, Huynh TK, Biering-Sorensen F. Return to work following spinal cord injury: a review. Disabil Rehabil. 2007 Sep 15;29(17):1341-75. doi: 10.1080/09638280701320839. PMID 17729082
- [Background] Marini, I., Lee, G. K., Chan, F., Chapin, M. H., & Romero, M. G. (2008). Vocational rehabilitation service patterns related to successful competitive employment outcomes of persons with spinal cord injury. Journal of Vocational Rehabilitation, 28(1), 1-13.
- [Background] O'Connor P. Incidence and patterns of spinal cord injury in Australia. Accid Anal Prev. 2002 Jul;34(4):405-15. doi: 10.1016/s0001-4575(01)00036-7. PMID 12067103
- [Background] Odendaal T. Injuries of the cervical spinal cord. The Ga-Rankuwa Hospital experience. S Afr Med J. 1991 Jul 20;80(2):75-9. PMID 1862438
- [Background] Odendaal T. Sub-cervical spinal injuries with neural involvement. The Ga-Rankuwa Hospital experience. S Afr Med J. 1991 Sep 7;80(5):219-23. PMID 1887346
- [Background] Office of the President (Office of the Status of Disbled People (South Africa). (1997). Integrated National Disability Strategy. Pretoria: Government Printer.
- [Background] Ottomanelli L, Lind L. Review of critical factors related to employment after spinal cord injury: implications for research and vocational services. J Spinal Cord Med. 2009;32(5):503-31. doi: 10.1080/10790268.2009.11754553. PMID 20025147
- [Background] Ottomanelli, L., Bradshaw, L.D.,Cipher, D.J. (2009). Employment and vocationl rehabilitation services use amogst veterans with spinal cord injury Journal of Vocational Rehabilitation, 31, 39-43.
- [Background] Ottomanelli L, Barnett SD, Goetz LL. Effectiveness of supported employment for veterans with spinal cord injury: 2-year results. Arch Phys Med Rehabil. 2014 Apr;95(4):784-90. doi: 10.1016/j.apmr.2013.11.012. Epub 2013 Dec 4. PMID 24316325
- [Background] Ottomanelli L, Barnett SD, Goetz LL. A prospective examination of the impact of a supported employment program and employment on health-related quality of life, handicap, and disability among Veterans with SCI. Qual Life Res. 2013 Oct;22(8):2133-41. doi: 10.1007/s11136-013-0353-5. Epub 2013 Jan 24. PMID 23345022
- [Background] Paddison, S. and Middleton, F. (2005). Physical Management in Neurological Rehabilitation. Third ed. Netherlands: Elsevier.
- [Background] Powell RA, Single HM. Focus groups. Int J Qual Health Care. 1996 Oct;8(5):499-504. doi: 10.1093/intqhc/8.5.499. PMID 9117204
- [Background] Faden RR, Powers M. Health inequities and social justice. The moral foundations of public health. Bundesgesundheitsblatt Gesundheitsforschung Gesundheitsschutz. 2008 Feb;51(2):151-7. doi: 10.1007/s00103-008-0443-7. PMID 18259708
- [Background] Ramakrishnan K, Mazlan M, Julia PE, Abdul Latif L. Return to work after spinal cord injury: factors related to time to first job. Spinal Cord. 2011 Aug;49(8):924-7. doi: 10.1038/sc.2011.16. Epub 2011 Mar 8. PMID 21383761
- [Background] Rabiee F. Focus-group interview and data analysis. Proc Nutr Soc. 2004 Nov;63(4):655-60. doi: 10.1079/pns2004399. PMID 15831139
- [Background] Raine,S.,Meadows.,Lynnch-Ellerington,M (2009). Bobath Concept: Theory and Clinical Practice in Neurological Rehabilitation.1st ed. West Sussex. Blackwell Publishing Ltd.
- [Background] Rankin G, Rushton A, Olver P, Moore A. Chartered Society of Physiotherapy's identification of national research priorities for physiotherapy using a modified Delphi technique. Physiotherapy. 2012 Sep;98(3):260-72. doi: 10.1016/j.physio.2012.03.002. Epub 2012 Apr 13. PMID 22898585
- [Background] Rauch A, Escorpizo R, Riddle DL, Eriks-Hoogland I, Stucki G, Cieza A. Using a case report of a patient with spinal cord injury to illustrate the application of the International Classification of Functioning, Disability and Health during multidisciplinary patient management. Phys Ther. 2010 Jul;90(7):1039-52. doi: 10.2522/ptj.20090327. Epub 2010 May 27. PMID 20508027
- [Background] Rauch A, Baumberger M, Moise FG, von Elm E, Reinhardt JD. Rehabilitation needs assessment in persons with spinal cord injury following the 2010 earthquake in Haiti: a pilot study using an ICF-based tool. J Rehabil Med. 2011 Nov;43(11):969-75. doi: 10.2340/16501977-0896. PMID 22031341
- [Background] Saulino, M. (2011). Rehabilitation of Persons With Spinal Cord Injuires. Medscape Reference. http://emedicine.medscape.com/article/1265209-overview#aw2aab6c12
- [Background] Schonherr MC, Groothoff JW, Mulder GA, Schoppen T, Eisma WH. Vocational reintegration following spinal cord injury: expectations, participation and interventions. Spinal Cord. 2004 Mar;42(3):177-84. doi: 10.1038/sj.sc.3101581. PMID 14758351
- [Background] Sinclair LB, Lingard LA, Mohabeer RN. What's so great about rehabilitation teams? An ethnographic study of interprofessional collaboration in a rehabilitation unit. Arch Phys Med Rehabil. 2009 Jul;90(7):1196-201. doi: 10.1016/j.apmr.2009.01.021. PMID 19577033
- [Background] Solagberu BA. Spinal cord injuries in Ilorin, Nigeria. West Afr J Med. 2002 Jul-Sep;21(3):230-2. doi: 10.4314/wajm.v21i3.28037. PMID 12744575
- [Background] Somers, M. (2001). Spinal Cord Injury: Functional Rehabilitation (2 ed.). New Jersey: Prentice Hall.
- [Background] South Africa. (1998). Employment Equity Act no 55 of 1998. Pretoria: Government Printer.
- [Background] South Africa. (2000). Promotion of Equality and Prevention of Unfair Descrimination Act no 4 of 2000. Pretoria: Government Printer.
- [Background] South Africa. (1995). Labour Relations Act no 66 of 1995. Pretoria: Government Printer.
- [Background] South Africa. (1998). Skills Development Act no 97 of 1998. Pretoria: Government Printer.
- [Background] South Africa. (1994). Public Service Act no 103 of 1994. Pretoria: Government Printer.
- [Background] South Africa. (1997). Basic Conditions of Employment Act no 11 of 1998. Pretoria: Government Printer.
- [Background] South Africa. (1996). Constitution of the Republic of South Africa no 108 of 1998. Pretoria: Government Printer.
- [Background] Stucki G. International Classification of Functioning, Disability, and Health (ICF): a promising framework and classification for rehabilitation medicine. Am J Phys Med Rehabil. 2005 Oct;84(10):733-40. doi: 10.1097/01.phm.0000179521.70639.83. No abstract available. PMID 16205428
- [Background] Targett P, Wehman P, Young C. Return to work for persons with spinal cord injury: designing work supports. NeuroRehabilitation. 2004;19(2):131-9. PMID 15201472
- [Background] Tomassen PC, Post MW, van Asbeck FW. Return to work after spinal cord injury. Spinal Cord. 2000 Jan;38(1):51-5. doi: 10.1038/sj.sc.3100948. PMID 10762198
- [Background] Umphred, D. (2007). Neurological Rehabilitation (5th ed.). St. Louis, Missouri: Mosby Elsevier.
- [Background] Vazquez-Ramos, R. L., M; Hernandez, NE. (2007). The Delphi Method in Rehabilitation Counselling Research Rehabilitation Counseling Bulletin, 50(2), 111-118.
- [Background] Velmahos GC, Degiannis E, Hart K, Souter I, Saadia R. Changing profiles in spinal cord injuries and risk factors influencing recovery after penetrating injuries. J Trauma. 1995 Mar;38(3):334-7. doi: 10.1097/00005373-199503000-00004. PMID 7897710
- [Background] Wilson, B., McLellan, D.L.(1997). Rehabilitation Studies Handbook.1st ed. Cambridge:Cambridge University Press.
- [Background] World Health Organisation. (2002).Towards a Common Language for Functioning, Disability and Health (ICF). Geneva: World Health Organization.
- [Background] Word Health Organisation (2013). International Perspectives on Spinal Cord Injury. Malta. World Health Organisation
- [Background] Zolna, J. S., J; Sabata, D; Goldthwaite, J. (2007). Review of accomodation strategies in the workplace for persons with mobility and dexterity impairments: Application to criteria for universal design Technology and Disability, 19, 189-198.
- [Derived] Pefile N, Mothabeng J, Naidoo S. A Multidisciplinary Model to Guide Employment Outcomes Among People Living With Spinal Cord Injuries in South Africa: A Mixed Methods Study Protocol. JMIR Res Protoc. 2016 Dec 6;5(4):e238. doi: 10.2196/resprot.5887. PMID 27923779